CLINICAL TRIAL: NCT00464243
Title: Efficacy and Safety of 2 mg/Day M100907 on Sleep Maintenance Insomnia: a 6-week, Multicenter, Randomized, Double-blind, Placebo-controlled Polysomnographic Study
Brief Title: Efficacy and Safety of Volinanserin on Sleep Maintenance Insomnia - Polysomnographic Study
Acronym: NOCTURNE907
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6072; EUDRACT : 2006-005303-34
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Sleep problems; Insomnia; Sleeplessness; Polysomnographic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — volinanserin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Volinanserin (Experimental): 2 mg volinanserin tablets orally once daily
  Interventions: Drug: volinanserin
- Placebo (Placebo Comparator): tablets orally once daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: volinanserin — oral administration
  Other Names: M100907
  Arms: Volinanserin
Drug: placebo — oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess efficacy and safety of volinanserin in the population of patients complaining of sleep maintenance insomnia. The patients suffering from that condition frequently wake up during the night, their sleep is non restorative and they suffer from a significant distress or impairment in their daily activities consecutive to insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary insomnia based on Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) criteria
* Disturbances of sleep maintenance criteria based on patient's information related to sleep pattern during the preceding month
* Specific criteria based on the NPSG recordings during the screening nights

Exclusion Criteria:

* Females who are lactating or who are pregnant
* Night shift workers, and individuals who nap 3 or more times per week over the preceding month
* Consumption of xanthine-containing beverages (i.e. tea, coffee, cola) comprising more than 5 cups/day
* Participation in another trial having received study medication within 1 month before the screening visit
* Body Mass Index ≥ 33
* Use of over-the-counter medications such as tryptophan, valerian root, kava, melatonin, St. John's Wort, Alluna or prescription sleep medication
* Use of any substance with psychotropic effects or properties know to affect sleep/wake
* History of primary hypersomnia, narcolepsy, breathing-related sleep disorder, circadian rhythm sleep disorder, parasomnia, dyssomnia
* Clinically significant, severe or unstable, acute or chronically progressive medical or surgical disorder
* Positive qualitative urine drug screen (opiates, cocaine, amphetamine…)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6 weeks of treatment of the mean night polysomnographic (NPSG) wake time after sleep onset (WASO). | 6 weeks

SECONDARY OUTCOMES:
Functional Outcomes of Sleep Questionnaire at 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Cove, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Laval, Quebec, Canada
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Moscow, Russia

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com